CLINICAL TRIAL: NCT02081833
Title: The Investigation of Methods to Capture Acute Respiratory and Gastrointestinal Infections of Children Aged 1 to 3 Years. Feasibility Study for the Braunschweig Birth Cohort LöwenKIDS (Infections and the Development of the Immune System)
Brief Title: The Investigation of Methods to Capture Acute Respiratory and Gastrointestinal Infections of Children Aged 1 to 3 Years
Status: Completed | Type: Observational
Sponsor: Helmholtz Centre for Infection Research (Other)
Responsible Party: Sponsor
Other Study IDs: 6506
Record Dates: First submitted 2014-02-28; First posted 2014-03-07 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Childhood Infections
Keywords: acute respiratory infections; acute gastrointestinal infections; children; child; symptom diary; nasal swabs; stool samples

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Parent-collected anterior-nasal swabs and stool samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Reminder group: the reminder group receives every 2 weeks a reminder to fill out the symptom diary (postcard or SMS)

SUMMARY:
This study serves as a feasibility study for a birth cohort study to investigate the influence of the sequence and load of infections and vaccinations on the development of the immune system of children. In this study, the investigators aim to test the methods developed to capture acute respiratory and gastrointestinal infections and their consequences of children aged 1 to 3 years in Braunschweig, Germany. Furthermore, the investigators want to study the influence of the environment on the microbiome of children by comparing children of the same child care centre with children from different child care centres. The methods developed include a symptom diary which has to be filled out on a daily basis by the parents. Furthermore parents are asked to take monthly anterior nasal swabs and stool samples from the study child independent from symptoms as well as one sample if symptoms occur. The parents are provided with instructions and the first nasal swab will be demonstrated by trained study personal. The study is powered to compare nasal swabs taken by the trained staff and the parents as primary outcome. Secondary outcome is the performance of reminders sent to the study participants. The diary and the specimen will be mailed to the Helmholtz Centre for Infection Research where they will be analyzed for the nasal and gut microbiome. The nasal swabs taken at the time of an infection will be tested for respiratory viruses. After the study period of 3 months parents will be asked about the feasibility and acceptance of the symptom diary and taking the nasal swabs and stool specimens by means of questionnaires and interviews (face to face and focus groups). This will help our understanding of the feasibility and acceptance of the methods developed to capture acute respiratory and gastrointestinal infections of children and our understanding of the development and composition of the nasal and gut microbiota.

DETAILED DESCRIPTION:
Further study details:

Recruitment takes place in child care centres (CCC) with children under the age of 3 years. In cooperation with the CCC, in the first step, the study is introduced to parents by leaflets and posters. In the second step, the study is personally introduced at the CCC with a brief presentation during an appointment or during the time parents pick up their child. Interested parents are handed out the consent forms and a first questionnaire with contact details to be sent back to the study team. After receipt of the signed informed consent, parents are contacted to schedule the appointment for the demonstration of the first nasal swab and for handing out the materials. From this day on, the 3-months study period starts for the parents. During these three months parents fill out the symptom diary on a daily basis and collect anterior nasal swabs and stool samples on a monthly basis from the study child independent from symptoms, as well as one sample if respiratory or gastrointestinal symptoms occur. 50% of the study participants are randomly chosen for the reminder subgroup; they receive 2-weekly reminders to continue the symptom diary by text messages or postcards.

The diary and the specimen will be mailed to the Helmholtz Centre for Infection Research where they will be stored and analyzed for the nasal and gut microbiome. The nasal swabs taken at the time of an infection will be tested for respiratory viruses, using a polymerase chain reaction (PCR) panel for 5 most common respiratory viruses (adeno-, influenza-, metapneumo-, picorna- and respiratory syncytial virus). All other nasal swabs will be tested for ß-actin and 16s rRNA as indicator for the quality of the nasal swab and the nasal swabs taken by the parents will then be compared with the nasal swabs taken by the trained study staff in a non-inferiority study.

After the study period of 3 months parents will be asked about the feasibility and acceptance of the tasks with questionnaires and interviews (face to face and focus groups).

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from both parents or legal guardians
* child below the age of three visiting a CCC in Braunschweig, Germany
* parents or guardian with sufficient German language skills to complete study diaries and perform study tasks as required

Exclusion Criteria:

* none

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children aged one to three years visiting a child care center in Braunschweig, Germany
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptance of taking nasal swabs and stool samples by parents of their child | after 3 months
  Feasibility and acceptance of taking nasal swabs and stool samples by parents of their child measured by:
  * the comparison of quality of nasal swab taken by trained study personal and swab taken by parents (ß-actin and 16s rRNA)
  * the number of samples sent back
  * the feedback by parents (by quantitative and qualitative methods)

SECONDARY OUTCOMES:
Composition of faecal and nasal microbiome | at baseline
  Similarity of the faecal and nasal microbiome among children from one child care centre

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Mikolajczyk, MD, MSc, Principal Investigator — Helmholtz Centre for Infection Research; André Karch, MD, MSc, Principal Investigator — Helmholtz Centre for Infection Research; Beate Zoch, MSc, Principal Investigator — Helmholtz Centre for Infection Research
Locations (1):
- Helmholtz Centre for Infection Research, Braunschweig, Lower Saxony, Germany